CLINICAL TRIAL: NCT01843088
Title: Randomized Trial of Mannitol Cream for Pain Relief After a Long Run
Brief Title: Trial of Mannitol Cream for Pain Relief After a Long Run
Acronym: PainCream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H13-00106
Record Dates: First submitted 2013-04-16; First posted 2013-04-30 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Pain
Keywords: Pain; exercise; muscle
MeSH Terms: conditions — Pain; Motor Activity | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mannitol cream (Experimental): cream containing 25% mannitol, applied as often and as much as needed to one leg ( chosen at random), on the day of a 10 km run, following the run and for five days afterwards
  Interventions: Drug: Mannitol cream
- Placebo cream (Placebo Comparator): Same carrier cream as that containing the active ingredient, mannitol, but without the active ingredient. Placebo cream to be applied to the painful areas of the other leg, chosen at random, on the day of a 10 km or more race, following the race, and as needed for the five days after the race. It is to be noted that, as almost no mannitol is absorbed through the skin, it is highly unlikely that this would involve the pain levels in the placebo leg.
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: Mannitol cream — 25% mannitol in PENcream (See above) (See above) This will be applied as needed to one side of the body (blinded assignment) over painful painful areas of legs following a 10 km run, on the day of the run and for five days afterwards.
  Other Names: Mannitol; PENcream, Commercially available proprietary cream.
  Arms: Mannitol cream
Drug: Placebo Cream — This is the vehicle only cream (PENcream) (See above) This will be applied as needed to one side of the body (blinded assignment) over painful painful areas of legs following a 10 km run, on the day of the run and for five days afterwards.
  Other Names: PENcream, commercially available proprietary cream.
  Arms: Placebo cream

SUMMARY:
Mannitol cream has been shown clinically to be effective for pain control. To determine if this effect is worth testing on a larger scale, 170 runners will receive a sample of 25% mannitol cream to apply on one leg, and the cream base without the mannitol on the other leg following a 10 km or longer run, and for the following five days. Mannitol and control legs will be chosen at random for each runner. Pain scores before and after cream application will be acquired each day for each leg. Means and standard deviations found will be used to determine the size of a larger study.

DETAILED DESCRIPTION:
The hypothesis for this study is that Mannitol cream will reduce post long run pain more than vehicle cream alone. In this parallel design, 170 runners who usually experience a pain level greater than 5/10 on a numerical rating scale from 0 to 10 where zero is no pain and 10 is the worst pain ever, will be given a cream containing 25% mannitol to apply on one leg and the vehicle cream to apply on the other leg. The cream assignment will be randomized, and the runner, the person supplying the cream and the person inputting the data will be blinded as to which leg received which cream. Pain levels in each leg following the long run will be recorded, via an e-mail questionnaire, or, failing this, by telephone, the day of the run, and each day, for five days following the run. Mean and standard deviations for pain levels will be calculated for each treatment leg, and a repeated measures ANOVA (Analysis Of VAriance) will be done comparing the pain levels in each leg over the six days. Using this information, if the NRS (Numeric rating scale) pain levels differ by more than 1/10 between the two groups, a larger study will be conducted using the information gathered in this study to determine sample size.

ELIGIBILITY:
Inclusion Criteria:

either:

* never ran 10 km or more, or;
* NRS pain level greater than 5/10 in both legs following a 10 km or more run

Exclusion Criteria:

* no major skin allergies
* no allergy to mannitol

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in NRS (Numeric rating scale) pain score | For six days following run
  NRS (Numeric rating scale) pain score from zero, no pain, to 10 worst pain ever. Change in pain score will be measured daily starting on day of race, comparing pain following the race, prior to the first cream application, to the daily scores for the subsequent five days. Pain levels in leg given mannitol cream, and leg given placebo cream will be compared according to the change in their pain scores.

SECONDARY OUTCOMES:
side effects of cream | For six days, starting on day of race.
  Description of side effects by subjects. The only likely to side effect would be a contact dermatitis as percutaneous systemic absorption of mannitol is negligible. We will therefore monitor for contact dermatitis, and record its incidence, should it happen in this small sample. In our experience with over 400 recipients, there have been no cases of contact dermatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Bertrand, MD, CCFP, Principal Investigator — University of British Columbia
Locations (1):
- Dr. Helene Bertrand, University of British Columbia, Department of Family Practice, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Cavone L, Calosi L, Cinci L, Moroni F, Chiarugi A. Topical mannitol reduces inflammatory edema in a rat model of arthritis. Pharmacology. 2012;89(1-2):18-21. doi: 10.1159/000335094. Epub 2012 Jan 10. PMID 22236612